CLINICAL TRIAL: NCT04789824
Title: The Impact of Eyelid Hygiene on Ocular Surface Among Opeartion Room Staff
Brief Title: The Impact of Eyelid Hygiene on Ocular Surface
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Aslı Nemli, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: surgerynurse
Record Dates: First submitted 2021-02-25; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Dry Eye
Keywords: dryeye; operation room; nurse; surgery; eyelid hygiene
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Single-blind, randomized-controlled
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigation group (Experimental): Eye Hygiene (warm compress, eyelid massage, and eyelid cleaning)
  Interventions: Behavioral: eyelid hygiene
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: eyelid hygiene — EH
  Arms: Investigation group

SUMMARY:
Dry eye is one of the most common eye diseases and it is known to be an ever-increasing public health problem in risky groups. Physical conditions (heat, light, humidity,ventilation), anesthetic gases, chemical-containing disinfectants and antiseptics are risk factors for dry eyes in operating rooms. In addition, the fact that surgery is a job that requires constant attention is considered among the factors that increase the risk of dry eye as it reduces the number of blinking. In the literature review, eye hygiene (hot application, massage, cleaning) is recommended as an application that protects and improves eye health. Because it has been reported to have significant positive effects on eye fatigue, dry eye symptoms and vision in both healthy and dry eyes. However, "daily eye hygiene" is a little-known practice in almost every society. In this context, the effect of eye hygiene on ocular surface moistening and vision-related quality of life in operating room workers was investigated in this study.The research was conducted as a randomized controlled experimental study between May 2018 and May 2019. All participants working in the operating room and meeting the inclusion criteria were included in the study. The group in which the participants will be included was determined by simple randomization. Eye hygiene training was given to the intervention group and eye hygiene practice was followed for 12 weeks. The control group was not intervened. Tear film stability and vision-related quality of life scores of both groups before and after 12 weeks of training were compared.

DETAILED DESCRIPTION:
Dry eye disease is one of the most common pathologies of the ocular surface which is characterized by tear film instability due to insufficient tear production or increased evaporation. Its prevalence varies between 5 to 50% in adults and may increase up to 75% in individuals aged above 40 years. This disease affects women twice as often as men. Dry eye poses burden on patients, due to associated symptoms that may widely range from persistent pain, itching, burning, stinging or scratchy and foreign body sensation, and light sensitivity to blurred vision, corneal epithelial defects, and ulcerations in the chronic state. In particular, in moderate-to-severe cases, pain, limitations in the daily living activities, and reduced quality of life are associated with depression, mood and sleep disorders. There are many factors proposed to play a role in the etiology of the disease: lifestyle habits, low humidity and artificial indoor heating and air conditioning systems, environmental factors such as air pollution containing chemical, physical, and biological pollutants, visual tasks requiring long-term mental focus, prolonged exposure to computer or smart phones, and occupational and personal habits that decrease the eyeblink frequency and increase the ocular evaporation.

The operating rooms are specially designed for multi-modality use and contain a number of environmental pollutants for the ocular surface associated with the physical environment and occupational and personal habits of healthcare providers. Surgery itself being a critical task demanding long-term mental focus, air conditioning, constant humidity, constant room temperature, intense lighting, irritant chemicals, surgical smoke, anesthetic gases, and biological aerosols are predisposing factors for ocular irritation in operating room staff. A few studies demonstrated that the risk of dry eye disease is higher in operating room staff, intensive care nursing and laboratory technicians. Castellanos-González et al. reported that their presence in the operating room predisposed surgical residents to have dry eye syndrome due to environmental conditions.

To the best of our knowledge, there is no study investigating the effectiveness of proper eyelid hygiene in dry eye disease among operating room staff., occupational activities with a high level of visual burden, and working environment. Dry eye disease is a chronic and progressive condition. Treatment provides symptomatic relief; however, cure is seen in only a small fraction of patients. The 2017 Tear Film and Ocular Surface Society (TFOS) revisited the management and treatment of dry eye disease in a two-step model. Accordingly, in the first step, non-pharmacological methods such as education about the disease and its management, modification of local environment, dietary changes, increasing fluid intake, enhanced blinking behavior, and proper eyelid hygiene are recommended. Based on these recommendations, eyelid hygiene regimen consisting of warm compress, lid massage, and eye cleaning is a supportive and rehabilitative approach. Also, studies have revealed that have also demonstrated the favorable effects of daily eyelid hygiene consisting of warm compress, lid massage, and cleaning on eye fatigue, dry eye symptoms, and visual acuity and recommended this regimen as a preventive medicine and health promotion. Warm compress and mechanical lid massage induce the meibomian secretion (i.e., the tear film lipid layer is mostly (90%) derived from the meibomian oil secreted by the meibomian glands), while eye cleaning provides protein/lipid deposits around the eyelashes and eyelids and eliminates microbial agents such as Staphylococci and Demodex spp.

Previous studies have confirmed the increased the secretion of meibomian lipids that are pathologically altered with warm compress, the outcomes may vary depending on the duration of application, degree of heat, and patient compliance. It have shown that the mean temperature ranges between 37.7±0.3 and 41.6±1.0°C and the ideal temperature is 40 to 45°C for warm compress. Once the meibomian secretions are liquefied with warm compress, the main goal of lid massage is to reduce the clogging of the meibomian gland and to maintain sufficient drainage of the tears. Following eyelid warming for minimum four min once or twice daily, medium-to-intense eyelid massage has been shown to induce expression of the meibomian gland secretions. With similar effects to mechanical finger massage, intense pulsed light to the eyelid, high-frequency electrotherapy, meibomian gland compressors, and eye massagers with heat-vibration have been also utilized in studies. Previous studies have confirmed that eye clean is an effective approach to prevent meibomian gland dysfunction (MGD) and Demodex mites. The most common used eye clean regimens include warm water in a washcloth, soaked cloths, cotton pads, or cotton tipped applicators, and gentle rubbing with baby shampoo, alone or combined.

In the present study, we, for the first time, aimed to evaluate the impact of eyelid hygiene on tear film stability, ocular symptoms, and vision-related quality of life among operating room staff with Stage ≥I dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Actively working in the operating room setting, aged ≤50 years, and having Stage ≥1 dry eye disease. In a clinical examination by the ophthalmologist, volunteers with TBUT <10, Schirmer test <5, OSDI score ≥ 13, MQ score> 14.5, cornea or conjunctiva> 1 staining and reporting at least one severe ocular symptom

Exclusion Criteria:

* Active eye infection requiring treatment, receiving antihypertensives, antihistamines, psychogenic or chemotherapeutic agents, thyroid replacement therapy, or estrogen, having autoimmune diseases such as Sjögren's syndrome, rheumatoid arthritis, diabetes, or multiple sclerosis, having a previous anterior segment surgery, wearing contact lenses, receiving treatment for dry eye disease within the past six months, receiving omega-3 or vitamin A supplements currently or within the past three months, pregnant or lactating women, and menopausal or postmenopausal women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Stage ≥1 dry eye disease | Weeks 0.-10.
  Volunteers with Tear Break-up Time <10, Schirmer-1 test <5, Oclar Surface Disease Index score ≥ 13, McMonnies Questionnaire> 14.5 and reporting at least one severe ocular symptom (pain, stinging, burning, stinging, itching, dryness) were considered to be at least first stage dry eye.
Visual Function | Weeks 0.-10.
  Visual Function Questionnaire score 0-100

CONTACTS AND LOCATIONS:
Overall Officials: Aslı Nemli, PhD, Study Director — Erciyes Üniversitesi
Locations (2):
- Turkey (Türkiye) (2):
  - Aslı Nemli, Kayseri, Talas
  - Erciyes Universitesi Hastanesi, Kayseri